CLINICAL TRIAL: NCT00152516
Title: A Multi-Center, Open-Label, Long-Term, Follow-Up Study Of the Safety And Efficacy Of Levetiracetam In Children With Partial Onset Seizures.
Brief Title: Long-Term, Follow-Up Study Of the Safety And Efficacy Of Levetiracetam In Children With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01148; EudraCT number:2004-000200-40
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2010-01-13 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy, Partial
Keywords: Partial Onset Seizures; levetiracetam; Epilepsy; Keppra
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental)
  Interventions: Drug: levetiracetam (LEV)

INTERVENTIONS:
Drug: levetiracetam (LEV) — Per protocol oral tablets or oral solution at 10 to 30mg/kg/day bid for 48 weeks, or approximately 52 weeks should a subject choose to discontinue levetiracetam (LEV) at the end of the maintenance period.
  Other Names: Keppra

SUMMARY:
To allow pediatric patients with partial onset seizures an opportunity to receive (as follow-up to studies N01009(NCT00105040)/N01103(NCT00175890) or by direct enrollment) open-label levetiracetam treatment, continue studying cognition and behavior in children, and continue collection of safety/efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with partial onset seizures, with 1 to 2 anti-epileptic drugs (AEDS), with participation in previous levetiracetam pediatric studies (N01009 or N01103) or direct enrollment, for whom levetiracetam treatment will be of possible benefit

Exclusion Criteria:

* Patients on a ketogenic diet
* Seizures too close together to accurately count
* Pseudoseizures
* Status epilepticus 1 month prior Visit 1
* Current diagnosis of Lennox-Gastaut Syndrome or epilepsy secondary to a progressing cerebral disease will be excluded from the study.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2004-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (84):
- United States (38):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Loxahatchee Groves, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Saint Paul, Minnesota
  - Lebanon, New Hampshire
  - Edison, New Jersey
  - Voorhees Township, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Galveston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (6):
  - Campinas
  - Curitiba
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - São Paulo
- Canada (3):
  - Vancouver, British Columbia
  - Thornhill, Ontario
  - Toronto, Ontario
- Czechia (2):
  - Brno
  - Prague
- France (3):
  - Lille
  - Paris
  - Strasbourg
- Germany (6):
  - Kehl, Kork
  - Berlin
  - Erlangen
  - Heidelberg
  - Jena
  - Kiel
- Budapest, Hungary
- India (5):
  - Hyderabad
  - Lucknow
  - Mahim Mumbai
  - Mumbai
  - Pune Maharashtra
- Italy (4):
  - Calambrone
  - Genoa
  - Milan
  - Roma
- Mexico City, Mexico
- Gdansk, Poland
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Târgu Mureş
- Russia (3):
  - Kalingrad
  - Moscow
  - Saint Petersburg
- South Africa (3):
  - Cape Town
  - Capitol Park
  - Johannesburg
- United Kingdom (3):
  - Bristol
  - Cardiff
  - London

REFERENCES:
- [Result] Pina-Garza JE, Schiemann-Delgado J, Yang H, Duncan B, Hadac J, Hunter SJ. Adjunctive levetiracetam in patients aged 1 month to <4 years with partial-onset seizures: subpopulation analysis of a prospective, open-label extension study of up to 48 weeks. Clin Ther. 2010 Oct;32(11):1935-50. doi: 10.1016/j.clinthera.2010.09.017. PMID 21095488
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 102 sites in 17 countries participated in the study, of which 85 sites in 16 countries enrolled subjects in the study. First subject enrolled: 23 October 2004, Last subject last visit: 24 June 2008
Pre-assignment Details: Protocol amendment C2 (August 7, 2006) allowed direct enrollment from India, Australia, and New Zealand bypassing the blinded feeder studies N01009 and N01103.
Groups:
- Levetiracetam: Oral tablets or oral solution at 10 to 30 mg/kg/day bid for 48 weeks, or approximately 52 weeks should a subject choose to discontinue levetiracetam (LEV) at the end of the maintenance period.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 255 (Subjects that were dispensed at least 1 dose of study medication)
Completed | 180 (Subjects ongoing until study close-out)
Not Completed | 75
Not completed — Adverse Event | 18
Not completed — Lack and Loss of Efficacy | 30
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 8
Not completed — Protocol Violation | 3
Not completed — Other: Mother Refused To Cooperate | 1
Not completed — Other: Given Commercial Drug in Error | 2
Not completed — Other: Parents Withdrew Consent | 2
Not completed — Other: Non-Compliance | 2
Not completed — Other: Primary Care Physician's Decision | 1
Not completed — Other: Moved Out Of State | 1
Not completed — Other: Underwent Surgery for Epilepsy | 1
Not completed — Other: Sz Worsening, Seeking 2nd Opinion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam
Number analyzed (Participants) | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 255
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.28 (4.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 139
Region of Enrollment [Number; unit: participants]
  United States | 123
  Russian Federation | 7
  Italy | 6
  United Kingdom | 2
  India | 20
  France | 7
  Czech Republic | 9
  Hungary | 4
  Mexico | 6
  Canada | 11
  Poland | 2
  Brazil | 29
  Belgium | 4
  Romania | 7
  South Africa | 7
  Germany | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change (Reduction) of Partial (Type I) Seizure Frequency Per Week From Baseline Over Time During Treatment Period.
Description: Positive changes from Baseline indicate an improvement (i.e., a reduction) in seizure frequency per week.
Time Frame: Up-titration/Conversion Period (2-8 weeks); Maintenance Period (2-8 weeks to 40-46 weeks)
Population: 255 subjects were Intention to Treat (ITT), i.e. all subjects with at least 1 dose of study medication. Of these 255 ITT subjects 4 were missing a baseline, 3 had a baseline of 0, and 1 was missing treatment period seizure data. The result was a sample size of 247. Of these 247 subjects 226 continued into the maintenance period.
Measure: Median (Inter-Quartile Range); unit: percent reduction in seizures Per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 247
percent reduction in seizures Per Week
  Up-titration/Conversion | 51.06 [-10.70 to 91.59]
  Maintenance | 68.87 [-3.60 to 96.61]

2. Secondary Outcome: Percentage Change (Reduction) of Total (Type I, II, III) Seizure Frequency Per Week From Baseline Over Time During Treatment Period.
Description: Positive changes from Baseline indicate an improvement (i.e., a reduction) in seizure frequency per week.
Time Frame: Up-titration/Conversion Period (2-8 weeks); Maintenance Period (2-8 weeks to 40-46 weeks)
Population: 255 subjects were Intention to Treat (ITT), i.e. all subjects with at least 1 dose of study medication. Of these 255 ITT subjects 4 were missing a baseline, 2 had a baseline of 0, and 1 was missing treatment period seizure data. The result was a sample size of 248. Of these 248 subjects 227 continued into the maintenance period.
Measure: Median (Inter-Quartile Range); unit: Percent Reduction in Seizures per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 248
Percent Reduction in Seizures per Week
  Up-titration/Conversion Period | 47.44 [-21.18 to 88.70]
  Maintenance Period | 66.02 [-3.98 to 95.00]

3. Secondary Outcome: Partial (Type I) Seizure Frequency Per Week Over Time During Treatment Period.
Time Frame: Up-titration/Conversion Period (2-8 weeks); Maintenance Period (2-8 weeks to 40-46 weeks)
Population: 255 subjects were Intention to Treat (ITT), i.e. all subjects with at least 1 dose of study medication. Of these 255 ITT subjects 1 was missing treatment period seizure data leaving a sample size of 254. Of these 254 subjects 233 continued into the maintenance period.
Measure: Median (Inter-Quartile Range); unit: Seizures Per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 254
Seizures Per Week
  Up-titration/Conversion Period | 2.85 [0.23 to 26.30]
  Maintenance Period | 1.49 [0.07 to 17.89]

4. Secondary Outcome: Total (Type I, II, III) Seizure Frequency Per Week Over Time During Treatment Period.
Time Frame: Up-titration/Conversion Period (2-8 weeks); Maintenance Period (2-8 weeks to 40-46 weeks)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Seizures Per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 254
Seizures Per Week
  Up-titration/Conversion Period | 3.15 [0.25 to 31.17]
  Maintenance Period | 1.91 [0.09 to 24.86]

5. Secondary Outcome: Change (Reduction) From Baseline in Partial (Type I) Seizure Frequency Per Week Over Time During Treatment Period
Description: Positive changes from Baseline indicate an improvement (i.e., a reduction) in seizure frequency per week.
Time Frame: Up-titration/Conversion Period (2-8 weeks); Maintenance Period (2-8 weeks to 40-46 weeks)
Population: 255 subjects were Intention to Treat (ITT), i.e. all subjects with at least 1 dose of study medication. Of these 255 ITT subjects 4 were missing a baseline and 1 was missing treatment period seizure data. The result was a sample size of 250. Of these 250 subjects 229 continued into the maintenance period.
Measure: Median (Inter-Quartile Range); unit: Seizures Per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 250
Seizures Per Week
  Up-titration/Conversion Period | 0.72 [-0.81 to 7.14]
  Maintenance Period | 0.93 [-0.33 to 8.99]

6. Secondary Outcome: Change (Reduction) From Baseline in Total (Type I, II, III) Seizure Frequency Per Week Over Time During Treatment Period
Description: Positive changes from Baseline indicate an improvement (i.e., a reduction) in seizure frequency per week.
Time Frame: Up-titration/Conversion Period (2-8 weeks); Maintenance Period (2-8 weeks to 40-46 weeks)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Seizures Per Week
Arm/Group | Levetiracetam
Number analyzed (Participants) | 250
Seizures Per Week
  Up-titration/Conversion Period | 0.69 [-0.89 to 7.84]
  Maintenance Period | 0.93 [-0.33 to 10.70]

7. Secondary Outcome: Partial Seizure (Type I) Responder Rate (Percent) During the Up-titration/Conversion Phase and by Visit During the Maintenance Phase
Description: The responder rate is defined as the number of responders. A responder is a patient with a 50% or greater change (reduction) in partial seizure frequency per week.
  Note: Rates were reported as percentages.
Time Frame: Up-titration (4 weeks); Maintenance Visits 3-4 (weeks 4-14, 6-15, or 8-16); Visits 4-5 (weeks 14-24, 15-24, or 16-24); Visits 5-6 (weeks 24-36); Visits 6-7 (weeks 36-48)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 247
Percentage of Participants
  Up-titration/Conversion (4 weeks) | 50.6
  Maintenance Visits 3-4 (weeks 4-14, 6-15, or 8-16) | 59.8
  Maint. Visits 4-5 (weeks 14-24, 15-24, or 16-24); | 65.5
  Maintenance Visits 5-6 (weeks 24-36) | 68.2
  Maintenance Visits 6-7 (weeks 36-48) | 71.8

8. Secondary Outcome: Partial Seizure (Type I) Maximum Seizure Free Interval (Percentage of Days Belonging to a Seizure Free Interval of 28 Days or More)
Description: For subjects with up to 24 weeks in the evaluation phase the denominator for each subject is their number of days in the evaluation phase.
Time Frame: Subjects with up to 24 weeks of exposure
Population: Intention to Treat (ITT) subjects with <= 24 Weeks of Exposure and treatment period seizure data
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Levetiracetam
Number analyzed (Participants) | 51
Percentage of Days | 0.00 [0.00 to 0.00]

9. Secondary Outcome: Partial Seizure (Type I) Maximum Seizure Free Interval (Percentage of Days Belonging to a Seizure Free Interval of 28 Days or More)
Description: For subjects with greater than 24 weeks in the evaluation phase the denominator for each subject is their number of days in the evaluation phase.
Time Frame: Subjects with greater than 24 weeks of exposure
Population: Intention to Treat (ITT) Subjects with > 24 Weeks of Exposure and treatment period seizure data
Measure: Median (Inter-Quartile Range); unit: Percentage of days
Arm/Group | Levetiracetam
Number analyzed (Participants) | 203
Percentage of days | 61.49 [0.00 to 94.07]

10. Secondary Outcome: Total Seizure (Type I, II, III) Maximum Seizure Free Interval (Percentage of Days Belonging to a Seizure Free Interval of 28 Days or More)
Description: as for outcome 8
Time Frame: Subjects with up to 24 weeks of exposure
Population: Intention to Treat (ITT) Subjects with <= 24 Weeks of Exposure and treatment period seizure data
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Levetiracetam
Number analyzed (Participants) | 51
Percentage of Days | 0.00 [0.00 to 0.00]

11. Secondary Outcome: Total Seizure (Type I, II, III) Maximum Seizure Free Interval (Percentage of Days Belonging to a Seizure Free Interval of 28 Days or More)
Description: as for outcome 9
Time Frame: Subjects with greater than 24 weeks of exposure
Population: Intention to Treat (ITT) subjects with > 24 weeks of exposure and treatment period seizure data
Measure: Median (Inter-Quartile Range); unit: Percentage of Days
Arm/Group | Levetiracetam
Number analyzed (Participants) | 203
Percentage of Days | 58.41 [0.00 to 93.81]

12. Secondary Outcome: Total Seizure (Type I, II, III) Continuously Seizure Free During the Maintenance Period
Description: The measure description is the product limit adjusted percent of subjects seizure free starting from the beginning of the Maintenance Period.
  The up-titration period is the up to 6 week period of increasing dose prior to the Maintenance Period. The Maintenance Period is the period of stable dosing, subsquent to the up-titration period, which could last from 42 to 48 weeks.
Time Frame: greater than or equal to 24 weeks, greater than or equal to 40 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 233
Percentage of Participants
  >= 24 Weeks | 16.5
  >= 40 Weeks | 14.7

13. Secondary Outcome: Percent of Subjects With Each Seizure Type During the Evaluation Period
Description: Type I Seizure is a partial onset Seizure (see International League Against Epilepsy definitions).
  Type II Seizure is a Generalized Seizure (see International League Against Epilepsy definitions).
  Type III Seizure is a Unknown Seizure Type (see International League Against Epilepsy definitions).
  A subject could experience more than one seizure type.
Time Frame: Evaluation period (48 weeks)
Population: 255 subjects were Intention to Treat (ITT), i.e. all subjects with at least 1 dose of study medication. Of these 255 ITT subjects 1 was missing treatment period seizure data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 254
Percentage of Participants
  Type I | 88.6
  Type II | 12.9
  Type III | 7.1

14. Secondary Outcome: Investigator Global Evaluation Scale
Description: There are 7 categories, 3 for improvement (Marked improvement, Moderate improvement, Slight improvement), 3 for worsening (Slight worsening, Moderate worsening, Marked worsening), and 1 for no change (No change).
Time Frame: End of Evaluation period (week 48 or at point of early discontinuation)
Population: Intention to Treat (ITT) subjects for whom the assessment was performed
Measure: Number; unit: Percentage of Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 222
Percentage of Participants
  Improved | 76.1
  No Change | 15.3
  Worsened | 8.6

15. Secondary Outcome: Parent/Guardian Global Evaluation Scale
Description: as for outcome 14
Time Frame: End of Evaluation period (week 48 or at point of early discontinuation)
Population: Intention to Treat (ITT) subjects for whom the assessment was performed
Measure: Number; unit: Percentage of Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 214
Percentage of Participants
  Improved | 75.7
  No Change | 12.6
  Worsened | 11.7

16. Secondary Outcome: Subject (>=8 Years Old) Global Evaluation Scale
Description: as for outcome 14
Time Frame: End of Evaluation period (week 48 or at point of early discontinuation)
Population: Intention to Treat (ITT) subjects >= 8 years old for whom the assessment was performed
Measure: Number; unit: Percentage of Participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 71
Percentage of Participants
  Improved | 78.9
  No Change | 15.5
  Worsened | 5.6

17. Secondary Outcome: Leiter-R Associated Memory (AM) Memory Screen Composite Score Change From Baseline to Visit 5 (Week 24) and Visit 7 (Week 48) (4 to 16 Year Olds)
Description: The Leiter-R AM battery has 10 subtests. The raw scores of the subtests are converted into scaled scores. Six composite scores are constructed from the 10 subtest scaled scores. The Memory Screen is one of them. It is composed of 2 subtests the Associated Pairs and Forward Memory. The sum of the Associated Pairs and Forward Memory subtest scaled scores are converted into a Memory composite score normally distributed with a mean and standard deviation of 100 (±15). Higher scores and positive changes from baseline are better. The range of the Memory Screen composite score is 44 to 155.
Time Frame: Baseline to Visit 5 (Week 24) and Visit 7 (Week 48)
Population: At baseline there were 98 subjects with valid Memory Screen composite scores (mean=85.5, standard deviation=18.7). Of these 98 subjects, 87 had valid scores at Visit 5 (week 24) and 80 at Visit 7 (week 48).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Levetiracetam
Number analyzed (Participants) | 87
Score on a scale
  Visit 5 (week 24) | 4.8 (12.6)
  Visit 7 (week 48) | 4.5 (15.3)

18. Secondary Outcome: Bayley Scale of Infant Development (BSID) II Mental Development Index Scores Classification Shift From Baseline at Visit 5 (Week 24) (1 Month to < 4 Year Olds)
Description: This score is obtained from a total raw score which is the sum of a battery of individual questions. It is adjusted for a child's age, has an expected mean of 100 and standard deviation of 15, and can be categorized as: (1) Accelerated Performance (>= 115), (2) Within Normal Limits (85-114), (3) Mildly Delayed Performance (70-84), and (4) Significantly Delayed Performance (<=69). Changes from baseline are then further categorized where 'Improved' is any positive category change, 'Stable' is no category change, and 'Worsened' is any negative category change, from baseline.
Time Frame: Visit 5 (Week 24)
Population: The Bayley Scale of Infant Development (BSID) II assessment was performed only at selected sites where a neuropsychologist was available. Both a valid baseline and Visit 5 (week 24) assessment had to be present.
Measure: Number; unit: Number of subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 30
Number of subjects
  Worsened | 5
  Stable | 21
  Improved | 4

19. Secondary Outcome: Bayley Scale of Infant Development (BSID) II Mental Development Index Scores Classification Shift From Baseline at Visit 7 (Week 48) (1 Month to < 4 Year Olds)
Description: as for outcome 18
Time Frame: Visit 7 (week 48)
Population: The Bayley Scale of Infant Development (BSID) II assessment was performed only at selected sites where a neuropsychologist was available. Both a valid baseline and Visit 7 (week 48) assessment had to be present.
Measure: Number; unit: Number of subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 25
Number of subjects
  Worsened | 7
  Stable | 17
  Improved | 1

20. Secondary Outcome: Bayley Scale of Infant Development (BSID) II Psychomotor Development Index Scores Classification Shift From Baseline at Visit 5 (Week 24) (1 Month to < 4 Year Old)
Description: as for outcome 18
Time Frame: Visit 5 (week 24)
Population: as for outcome 18
Measure: Number; unit: Number of subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 29
Number of subjects
  Worsened | 1
  Stable | 20
  Improved | 8

21. Secondary Outcome: Bayley Scale of Infant Development (BSID) II Psychomotor Development Index Scores Classification Shift From Baseline at Visit 7 (Week 48) (1 Month to < 4 Year Old)
Description: as for outcome 18
Time Frame: Visit 7 (week 48)
Population: as for outcome 19
Measure: Number; unit: Number of subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 24
Number of subjects
  Worsened | 1
  Stable | 15
  Improved | 8

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 46/255
Other Adverse Events (participants affected / at risk) | 206/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=255)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hip dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Hepatic enzyme increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 5 (5)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1)
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 18 (22)
Infantile spasms (Nervous system disorders) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 6 (14)
Crying (Psychiatric disorders) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Oesophagogastric fundoplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=255)
Constipation (Gastrointestinal disorders) | 18 (24)
Diarrhoea (Gastrointestinal disorders) | 34 (45)
Vomiting (Gastrointestinal disorders) | 41 (62)
Irritability (General disorders) | 27 (33)
Pyrexia (General disorders) | 81 (131)
Bronchitis (Infections and infestations) | 16 (22)
Ear infection (Infections and infestations) | 18 (29)
Influenza (Infections and infestations) | 16 (22)
Nasopharyngitis (Infections and infestations) | 38 (53)
Otitis media (Infections and infestations) | 21 (34)
Pharyngitis (Infections and infestations) | 15 (30)
Rhinitis (Infections and infestations) | 14 (20)
Upper respiratory tract infection (Infections and infestations) | 62 (105)
Somnolence (Nervous system disorders) | 20 (24)
Decreased appetite (Metabolism and nutrition disorders) | 14 (17)
Convulsion (Nervous system disorders) | 17 (20)
Headache (Nervous system disorders) | 31 (46)
Aggression (Psychiatric disorders) | 15 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (39)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (20)
Rash (Skin and subcutaneous tissue disorders) | 24 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.